CLINICAL TRIAL: NCT02657070
Title: Desaprendiendo la parálisis Aprendida Con RGS en Pacientes Afectos de Ictus
Brief Title: Counteracting Learned Non-use Through Augmented Visuomotor Feedback in Virtual Reality (RGS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Pompeu Fabra (Other)
Collaborators: Hospital Universitari Joan XXIII de Tarragona. (Other)
Responsible Party: Principal Investigator, Paul Verschure, Prof., Universitat Pompeu Fabra
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEIC 53/2013
Record Dates: First submitted 2016-01-13; First posted 2016-01-15 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Hemiparesis
Keywords: Stroke; learned non-use; Virtual Reality; Hemiparesis
MeSH Terms: conditions — Paresis; Stroke | interventions — PITX2 protein, human

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Experimental Group (Experimental): Virtual reality based therapy with augmented visuomotor feedback.
  Interventions: Behavioral: Reinforcement-Induced Movement Therapy (RIMT)
- Control Group (Active Comparator): Virtual reality based therapy without augmentation.
  Interventions: Behavioral: VR-based motor rehabilitation in RGS without augmented feedback

INTERVENTIONS:
Behavioral: Reinforcement-Induced Movement Therapy (RIMT) — 6 weeks, 1 session a day, 30min per sessions, of physical therapy using a VR rehabilitation gaming system (RGS) with augmented visuomotor feedback
  Other Names: VR-based motor rehabilitation in RGS with amplified visuomotor feedback
  Arms: Experimental Group
Behavioral: VR-based motor rehabilitation in RGS without augmented feedback — 6 weeks, 1 session a day, 30min per sessions, of physical therapy using a VR rehabilitation gaming system (RGS)
  Arms: Control Group

SUMMARY:
The purpose of this study is to determine if Reinforcement-Induced Movement Therapy (RIMT), a novel rehabilitation method that augments visuomotor feedback of movements of the patient in virtual reality, is effective in treating hemiparesis resp. learned non-use.

ELIGIBILITY:
Inclusion Criteria:

* Mild-to-moderate upper-limbs hemiparesis (Proximal Medical Research Council Scale > 2) due to ischemic or hemorrhagic stroke
* Spasticity in the affected limb (Modified Ashworth Scale <3)
* First-ever ischemic or hemorrhagic stroke (>4 weeks post-stroke)
* Sufficient cognitive capacity for following the instruction of the intervention (Mini-Mental State Evaluation >24)

Exclusion Criteria:

* Cognitive impairment that impede the correct execution or understanding of the intervention
* Severe impairments in vision or visual perception abilities (such as vision loss or spatial neglect), in spasticity, in communication abilities (such as aphasia or apraxia), severe pain as well as other neuromuscular or orthopedic changes that impede the correct execution of the intervention training
* Mental dysfunctioning during the acute or subacute phase after the stroke.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The upper extremity Fugl-Meyer Assessment | at baseline, at 6-weeks (after intervention), and at 12-weeks follow-up
  change from baseline in motor function

SECONDARY OUTCOMES:
Chedoke Arm Hand Inventory | at baseline, at 6-weeks (after intervention), and at 12-weeks follow-up
  change from baseline in functional recovery
Barthel Index | at baseline, at 6-weeks (after intervention), and at 12-weeks follow-up
  change from baseline in activities of daily living
Hamilton Scale | at baseline, at 6-weeks (after intervention), and at 12-weeks follow-up
  change from baseline in measurement of depression

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Maria San Segundo Mozo, Dra., Principal Investigator — Medico Especialista en Medician Fisica y Rehabilitation, Doctora por al Universitat Rovira i Virgili de Tarragona; Paul F.M.J. Verschure, Prof., Study Director — Director SPECS

REFERENCES:
- [Background] Ramachandran VS, Rogers-Ramachandran D. Phantom limbs and neural plasticity. Arch Neurol. 2000 Mar;57(3):317-20. doi: 10.1001/archneur.57.3.317. PMID 10714655
- [Background] de Haan RJ, Limburg M, Van der Meulen JH, Jacobs HM, Aaronson NK. Quality of life after stroke. Impact of stroke type and lesion location. Stroke. 1995 Mar;26(3):402-8. doi: 10.1161/01.str.26.3.402. PMID 7886714
- [Background] Thomas SA, Lincoln NB. Factors relating to depression after stroke. Br J Clin Psychol. 2006 Mar;45(Pt 1):49-61. doi: 10.1348/014466505X34183. PMID 16480566
- [Background] Robinson RG, Jorge RE. Post-Stroke Depression: A Review. Am J Psychiatry. 2016 Mar 1;173(3):221-31. doi: 10.1176/appi.ajp.2015.15030363. Epub 2015 Dec 18. PMID 26684921
- [Derived] Ballester BR, Maier M, San Segundo Mozo RM, Castaneda V, Duff A, M J Verschure PF. Counteracting learned non-use in chronic stroke patients with reinforcement-induced movement therapy. J Neuroeng Rehabil. 2016 Aug 9;13(1):74. doi: 10.1186/s12984-016-0178-x. PMID 27506203